CLINICAL TRIAL: NCT01913145
Title: Usability and HbA1c Method Comparison Study Using Lay Person Micro-Blood Specimens
Brief Title: Comparison Study of Lay Person Finger Stick Versus Blood Draw
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Home Access Health Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 040412
Record Dates: First submitted 2013-03-21; First posted 2013-07-31 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A1c, Self-collection, Blood sample (Experimental): Can a lay-persons safely and effectively self-collect a capillary blood sample of sufficient adequacy for A1c ("HbA1c") testing in a clinical laboratory
  Interventions: Device: A1c, Self-collection, Blood sample

INTERVENTIONS:
Device: A1c, Self-collection, Blood sample — This is a study to evaluate the safety and effectiveness of Micro-Serum/Micro-Blood (finger Stick) Specimen Collection as compared to samples obtained by standard venipuncture (blood taken from the arm vein).
  Other Names: HomeAccess A1c Kit

SUMMARY:
This is a study to evaluate the safety and effectiveness of Micro-Serum/Micro-Blood (finger Stick) Specimen Collection as compared to samples obtained by standard venipuncture (blood taken from the arm vein).

DETAILED DESCRIPTION:
This is a study to evaluate the safety and effectiveness of Micro-Serum/Micro-Blood (finger Stick) Specimen Collection as compared to samples obtained by standard venipuncture (blood taken from the arm vein). The information and data obtained will be used to finish development of a convenience kit that allows doctors to provide their patients a method to have their blood tested for clinical laboratory tests in the convenience of their home without having to visit the doctor's office or clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and follow verbal and written instructions in English
2. Demonstrate a willingness to participate by providing a written informed consent
3. Aged between 18 to 80 years of age with no obvious signs of illness (e.g. fever, vomiting)
4. Diabetics who were diagnosed 6 months ago or longer are preferred. However, non-diabetics will be accepted into the study.

Exclusion Criteria:

1. Withdrawn informed consent
2. Mental or physical impairment which would preclude participation
3. Any condition which, in the opinion of the Principle Investigator or site or study coordinator, makes the participant unsuitable for this study. This includes but is not limited to any mental or physical impairment, which would preclude provision of adequate and knowledgeable consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Usability and HbA1c Method Comparison Study Using Lay-Person Micro-Blood Specimens | Outpoint measured within 3 months
  To establish that when using capillary blood collected in the Home Access Collection Cassette, lay-users can obtain HbA1c results equivalent to results from professionally-collected samples

CONTACTS AND LOCATIONS:
Overall Officials: David Klonoff, MD, Principal Investigator — Mills-Peninsula Health Services Dorothy L. and James E. Frank Diabetes Research Institute 100 South San Mateo Drive San Mateo, California 94401; Harold E. Bayes, MD, Principal Investigator — L-MARC, 3288 Illinois Ave., Louisville, KY
Locations (2):
- United States (2):
  - Mills-Peninsula Health Services, San Mateo, California
  - L-MARC, Louisville, Kentucky